CLINICAL TRIAL: NCT04379388
Title: Improving Smoking Cessation in Socioeconomically-Disadvantaged Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Andrea Villanti, Associate Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-0351; P20GM103644 (NIH)
Record Dates: First submitted 2020-04-24; First posted 2020-05-07 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Nicotine Dependence, Cigarettes
Keywords: smoking; smoking cessation; nicotine; nicotine dependence
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web + text smoking cessation intervention (Experimental): Participants will receive referral to a quit smoking hotline and 12-week web and text-based smoking cessation intervention
  Interventions: Behavioral: Web + text smoking cessation intervention
- Usual care control (No Intervention): Participants will receive referral to a quit smoking hotline

INTERVENTIONS:
Behavioral: Web + text smoking cessation intervention — Participants will receive referral to a quit smoking hotline and 12-week web and text-based smoking cessation intervention
  Arms: Web + text smoking cessation intervention

SUMMARY:
The purpose of this study is to understand how to develop and deliver a better smoking cessation program for lower-income young adult smokers.

DETAILED DESCRIPTION:
Using content and strategy developed from the formative research phase, this randomized smoking cessation trial will test the impact of a tailored cessation intervention for socioeconomically-disadvantaged young adult (SDYA) smokers compared to a usual-care control on intervention engagement, self-efficacy to quit, and 30-day point prevalence abstinence at 3-month follow-up.

This study will take place over a 3-month period. Individuals who complete the screening survey and are eligible to participate will be asked to complete a 15-20 minute baseline survey at the start of the study. This survey will ask questions about use of mobile phones, tobacco use, recent alcohol and other drug use, concerns about the coronavirus outbreak and how it may affect personal tobacco use, and physical activity. After the first survey, participants will be assigned randomly to one of two study groups:

Group A: Referral to a quit smoking hotline (quit line)

Group B: Referral to a quit smoking hotline (quit line), plus enrollment in a web and text-based smoking cessation intervention.

Participants in both groups will be enrolled after completing the following steps, in order:

1. Providing consent to participate in the study;
2. Confirming contact information;
3. Completing a payment acknowledgement form that allows us to reimburse for survey/task completions; and
4. Completing the baseline survey.

To complete enrollment, participants in Group B will also be required to register for an account on BecomeAnEx.org and enroll in text messages on the site. Once registered, Group B participants will be enrolled in a text message program customized for this study and will need to respond to the initial message from the text message platform to initiate text messages.

Participants in Group B will receive daily text messages for 3 months with content delivered through the Truth Initiative's BecomeAnEx digital quit smoking platform. They will also receive brief (1-2 minute) weekly check-in surveys related to the week's messages and smoking status during this time.

At 3-months, participants in both groups will receive the 15-minute follow-up assessment. Participants in both groups who report quitting smoking at 3-months will be mailed a kit in order to take a saliva test to measure the amount of cotinine, a metabolite of nicotine, in their saliva. Participants who report smoking at the 3-month follow-up will not receive this saliva test.

All study procedures will take place remotely, with surveys conducted online. Participants in Group A will be paid at least $30 for participation and up to $80. Participants in Group B will be paid at least $40 for participation and up to $170.

ELIGIBILITY:
Inclusion Criteria:

* age 18-30
* lives in the U.S.
* smoked at least 100 lifetime cigarettes
* currently smokes every day or some days
* interest in quitting smoking within the next 6 months
* subjective financial situation of just meeting or not meeting basic expenses
* access to a smartphone with internet

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 437 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
30-day point prevalence smoking abstinence | Assessed at 3-month follow-up
  Self-reported smoking abstinence and biochemical validation (saliva cotinine)
Self-efficacy to quit smoking | Assessed at 3-month follow-up
  Confidence to quit within the next month (7days) on 0-10 scale
Intervention engagement | 12 weeks
  Completing 75% or more of 12 weekly check-ins

SECONDARY OUTCOMES:
7-day point prevalence smoking abstinence | Assessed at 3-month follow-up
  Self-reported smoking abstinence
Number of 24-hour quit attempts | Assessed at 3-month follow-up
  Number of times intentionally stopped smoking cigarettes for 24 hours or longer because trying to quit
Perceived support to quit smoking | Assessed 3-month follow-up
  4 items pertaining to quit support from the text messages
Pattern and rate of tobacco/e-cigarette use | Assessed at 3-month follow-up
  Past 30 (90 day) use of tobacco or nicotine products such as cigars, e-cigarettes, chewing tobacco, and nicotine replacement products

CONTACTS AND LOCATIONS:
Overall Officials: Andrea C Villanti, PhD, MPH, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No